CLINICAL TRIAL: NCT04668404
Title: Study of Coagulation Profile and Role of Heparin-like Effect in Patients With COVID-19
Brief Title: Study of Coagulation Profile and Role of Heparin Like Effect in Patients With COVID-19
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, KAMAL KAJAL, ASSOCIATE PROFESSOR, DEPT. OF ANAESTHESIA AND INTENSIVE CARE,, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IEC-04/2020-1641
Record Dates: First submitted 2020-12-10; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Hypercoagulable States Nec
Keywords: COVID-19; Sonoclot; hypercoagulable; ARDS
MeSH Terms: conditions — COVID-19; Thrombophilia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 positive patient with ARDS: All patients with COVID-19 diagnosed with RT-PCR.
  Interventions: Diagnostic Test: Sonoclot

INTERVENTIONS:
Diagnostic Test: Sonoclot — Sonoclot machine

SUMMARY:
Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection is a pandemic, which has affected approximately 4 lakhs individuals and claimed 16,362 deaths till now. SARS-CoV-2 has been associated with myocarditis and renal dysfunction. Patients hospitalized for Covid-19 severe infection are more prone to excessive coagulation activation leading to thrombotic events both in the venous and arterial circulations, due to excessive inflammation, platelet activation, endothelial dysfunction, and stasis. Nearly 20% of COVID-19 patients present severe coagulation abnormalities, which may occur in almost all of the severe and critical ill COVID-19 cases. Concomitant venous thromboembolism (VTE), a potential cause of unexplained deaths, has been frequently reported in COVID-19 cases, but its management is still challenging due to the complexity between antithrombotic therapy and coagulation disorders. The importance of high D-dimer and Fibrin degradation product level to determine the patient prognostic and the risk of thrombosis is known. In a French study, it was found that a high rate of thromboembolic events in COVID-19 patients treated with therapeutic anticoagulation, with 56% of VTE and 6 pulmonary embolisms. Preliminary reports on COVID-19 patients' clinical and laboratory findings include thrombocytopenia, elevated D-dimer, prolonged prothrombin time, and disseminated intravascular coagulation. COVID-19 patients with acute respiratory failure present a severe hypercoagulability rather than consumptive coagulopathy.

Another study highlights this common finding in most COVID-19 patients with high D-dimer levels which are associated with a worse prognosis. Cases showed significantly higher fibrinogen and D-dimer plasma levels versus healthy controls (p < 0.0001). Markedly hypercoagulable thromboelastometry profiles were observed in COVID-19 patients, as reflected by shorter Clot Formation Time (CFT) in INTEM (p = 0.0002) and EXTEM (p = 0.01) and higher Maximum Clot Firmness (MCF). Fibrin formation and polymerization may predispose to thrombosis and correlate with a worse outcome.

Global VE tests provide a more physiologic assessment of coagulation and should be considered to guide blood transfusion requirements in liver transplantation and other major surgery. Its application in patients with Covid19 or in a critical care setting requires more data. Viscoelastic tests, which include TEG, ROTEM, and Sonoclot, offer a means of assessing the activity of pro-and anticoagulant pathways, hyperfibrinolysis, and excessive clot lysis. Assessment of clot formation can be performed in 10 to 20 minutes as a point of care (POC) test; however, assessment of clot lysis takes 30 to 60 minutes. SIRS and sepsis trigger the release of endogenous heparinoids, or a heparin-like effect (HLE), due to small endothelium/mast cell-derived glycosaminoglycan's, which can be detected on heparinase-treated viscoelastic assays.

Viscoelastic testing of global coagulation such as thromboelastometry and Sonoclot has been proposed as a superior tool to rapidly diagnose and help guide resuscitation with blood products and anticoagulation. it is deemed necessary to determine the influence of Covid 19 on coagulation parameters using point of care coagulation using sonoclot and conventional coagulation tests. In this prospective trial, the investigators aim to evaluate coagulation abnormalities via traditional tests and whole blood Sonclot profiles in a group of 50 consecutive patients with critically ill COVID-19 patients admitted to the Covid ICU OF Nehru Hospital extension, Postgraduate Institute of Medical Education and Research, Chandigarh.

DETAILED DESCRIPTION:
Several Consensus statements have been published in the literature in the last 2 months emphasizing the need for data in Covid 19 to assess the risk of both bleeding i.e. disseminated intravascular coagulation (DIC) and thromboses (stoke, myocardial infarction, dialysis catheter blocks).

Early reports showed that very high D-dimer levels are common in COVID-19 pneumonia and correlate with a worse prognosis. To better characterize COVID-19-related coagulation changes, many studies are showing some initial data regarding the role of procoagulant micro thrombotic changes rather than DIC. Coagulation profiles observed in studies published in the last one month reflect a severe hypercoagulability rather than a consumptive coagulopathy (e.g., disseminated intravascular coagulation). Such a laboratory pattern and association can be linked to both markedly increased levels of fibrinogen and an excessive fibrin polymerization due to the infection. SARS-CoV-2 is likely to promote massive fibrin formation and deposition which can also account for the extremely high D-dimer levels found in these patients. Fibrin deposition in alveolar and interstitial lung spaces, in addition to microcirculation thrombosis, may contribute to worsening respiratory failure resulting in prolonged mechanical ventilation, poor prognosis, and death. Furthermore, other major venous thromboembolic events and arterial complications (e.g., acute myocardial infarction) have been reported and are likely to be largely underestimated. In this regard, anticoagulant therapy may improve the prognosis in COVID19 patients as reported by various studies. In light of the severe hypercoagulable state observed in these patients, effective anticoagulant prophylaxis should be considered to reduce the risk of thrombotic complications. This will be the first prospective study to assess the impact of adequate dosages of anticoagulants on clotting parameters in an Indian scenario.

There are several ways in which the COVID-19 pandemic may affect the prevention and management of the thrombotic and thromboembolic disease.

* First, the direct effects of COVID-19 or the indirect effects of infection, such as through severe illness and hypoxia, may predispose patients to thrombotic events. Preliminary reports suggest that hemostatic abnormalities, including disseminated intravascular coagulation (DIC), occur in patients affected by COVID-19.
* Additionally, the severe inflammatory response, critical illness, and underlying traditional risk factors may all predispose to thrombotic events, similar to prior virulent zoonotic coronavirus outbreaks.
* Investigational therapies for treating COVID-19 may have adverse drug-drug interactions with antiplatelet agents and anticoagulants.
* Lastly the pandemic, because of resource allocations or social distancing recommendations, may adversely affect the care of patients without COVID-19 but who present with thrombotic events. For example, (mis)perception that antithrombotic agents confer increased risk for contracting COVID-19, may lead to untoward interruption of anticoagulation by some patients

Further, a few of these investigational agents being used for Covid19 have been associated with excess risk (or, in other cases, reduced risk) for thrombotic events, or for thrombocytopenia in prior studies of non-COVID-19 populations. For example, bevacizumab, a monoclonal antibody that binds to vascular endothelial growth factor (VEGF), and is under investigational use for COVID-19, is associated with increased risk for adverse cardiovascular events, including MI, cerebrovascular accidents, and venous thromboembolism (VTE). Alternatively, fingolimod, an immunomodulating agent being tried for COVID-19, may reduce reperfusion injury and improve outcomes in patients suffering from acute ischemic stroke. Hydroxychorloquine, recently receiving Emergency Use Authorization from the U.S. Food and Drug Administration for treatment of COVID-19, may potentially exert antithrombotic properties, especially against anti-phospholipid antibodies.

There is no data available on the subject of India. However preliminary data from our institute suggest the following which is in concordance with published data elsewhere

* The most consistent hemostatic abnormalities with COVID-19 include mild thrombocytopenia and increased D-dimer levels, which are associated with a higher risk of requiring mechanical ventilation, intensive care unit [ICU] admission, or death.
* Disease severity is variably associated with prolongation of the prothrombin time (PT) and international normalized ratio (INR) and variably by a trend toward shortened activated partial thromboplastin time (aPTT).

Hospitalized patients with COVID-19 who have respiratory failure or co-morbidities (e.g., active cancer, or heart failure), patients who are bedridden, and those requiring intensive care should receive pharmacological VTE prophylaxis, unless there are contraindications. The choice of agents and dosing should be based on available guideline recommendations. The World Health Organization interim guidance statement recommends prophylactic daily low-molecular weight heparins (LMWHs), or twice daily subcutaneous unfractionated heparin (UFH). If pharmacological prophylaxis is contraindicated, mechanical VTE prophylaxis (intermittent pneumatic compression) should be considered in immobilized patients. In this regard, the once-daily dosing regimen of LMWHs may be advantageous over UFH to reduce personal protective equipment (PPE) use and exposure of healthcare workers.

POC test services as quality assured pathology services using analytical devices (including test kits and analysers), provided near to the patient rather than in the traditional environment of a clinical laboratory.

These POC tests can be classified as Viscoelastic POC (vPOC) tests which include Thromboelastography (TEG), rotation thromboelastometry (ROTEM), and Sonoclot; and Platelet function tests which are Platelet function analyser, etc. TEG, ROTEM, and Sonoclot analysis are point-of-care coagulation monitoring devices which assess the viscoelastic properties of whole blood. They measure the entire clotting process, at the bedside and in a sample of whole blood. Coagulation factors present in plasma interact with platelets and red cells displaying results in a pictorial manner starting with fibrin formation and continue through clot retraction and fibrinolysis.

The role of SCTS for coagulation correction in patients with Covid19 is unclear and using POC tests in ICUs will be of great help in tailoring treatment

Investigators will also try to determine the influence of sepsis on coagulation disorders in COVID - 19 patients, to correctly identify the type and optimal quantity of blood product requirement in at-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Age 18-80 years
  * Confirmed Covid19 patient with positive RT PCR
* Exclusion Criteria:

  * Current therapy: Recent blood or blood component transfusion in the last 2 weeks.
  * HIV positive/ AIDS patients
  * Pregnancy
  * Active malignancy within the last 5 years
  * Not willing to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with COVID-19 admitted in ICU/ HDU, admitted under the department of medicine and anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of of conventional coagulation tests with point of care coagulation test using sonoclot in COVID-19 patients. | 1 month
  To correlate conventional coagulation tests with point of care coagulation test using sonoclot

SECONDARY OUTCOMES:
Clinical Evidence of thrombosis | 1 month
  Coagulation Related Thromboembolic events
Coagulation-related Bleeding Event | 28 days
  Coagulation-related Bleeding Event
Presence of Endogenous Heparinoids as demonstrated on POC test [ Time Frame 0, 3 days] | [ Time Frame 0, 3 days
  Presence of Endogenous Heparinoids as demonstrated on POC test [ Time Frame 0, 3 days]
Intensive care admission duration | 28 days
  Intensive care admission duration
28 day mortality | 28 days
  28 day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sukriti S, Maras JS, Bihari C, Das S, Vyas AK, Sharma S, Hussain S, Shasthry S, Choudhary A, Premkumar M, Kumar D, Kumar G, Mukhopadhyay C, Kumar A, Trehanpati N, Rautou PE, Moreau R, Sarin SK. Microvesicles in hepatic and peripheral vein can predict nonresponse to corticosteroid therapy in severe alcoholic hepatitis. Aliment Pharmacol Ther. 2018 Apr;47(8):1151-1161. doi: 10.1111/apt.14564. Epub 2018 Feb 20. PMID 29460445
- [Result] Premkumar M, Bihari C, Saxena P, Devurgowda DR, Vyas T, Mirza R, Jain P, Kumar G, Bhatia P, Baweja S, Choudhury A, Sarin SK. Heparin-like Effect Associated With Risk of Bleeding, Sepsis, and Death in Patients With Severe Alcohol-Associated Hepatitis. Clin Gastroenterol Hepatol. 2020 Feb;18(2):486-495.e3. doi: 10.1016/j.cgh.2019.04.057. Epub 2019 May 8. PMID 31077821
- [Result] Premkumar M, Devurgowda D, Dudha S, Maiwall R, Bihari C, Grover S, Gupta E, Kumar S, Sarin SK. A/H1N1/09 Influenza is Associated With High Mortality in Liver Cirrhosis. J Clin Exp Hepatol. 2019 Mar-Apr;9(2):162-170. doi: 10.1016/j.jceh.2018.04.006. Epub 2018 May 17. PMID 31024197
- [Result] Premkumar M, Rangegowda D, Kajal K, Khumuckham JS. Noninvasive estimation of intravascular volume status in cirrhosis by dynamic size and collapsibility indices of the inferior vena cava using bedside echocardiography. JGH Open. 2019 Mar 12;3(4):322-328. doi: 10.1002/jgh3.12166. eCollection 2019 Aug. PMID 31406926
- [Result] Harzallah I, Debliquis A, Drenou B. Lupus anticoagulant is frequent in patients with Covid-19. J Thromb Haemost. 2020 Aug;18(8):2064-2065. doi: 10.1111/jth.14867. Epub 2020 May 11. No abstract available. PMID 32324958
- [Result] Panigada M, Bottino N, Tagliabue P, Grasselli G, Novembrino C, Chantarangkul V, Pesenti A, Peyvandi F, Tripodi A. Hypercoagulability of COVID-19 patients in intensive care unit: A report of thromboelastography findings and other parameters of hemostasis. J Thromb Haemost. 2020 Jul;18(7):1738-1742. doi: 10.1111/jth.14850. Epub 2020 Jun 24. PMID 32302438
- [Result] Lippi G, Plebani M, Henry BM. Thrombocytopenia is associated with severe coronavirus disease 2019 (COVID-19) infections: A meta-analysis. Clin Chim Acta. 2020 Jul;506:145-148. doi: 10.1016/j.cca.2020.03.022. Epub 2020 Mar 13. PMID 32178975
- [Result] Intagliata NM, Argo CK, Stine JG, Lisman T, Caldwell SH, Violi F; faculty of the 7th International Coagulation in Liver Disease. Concepts and Controversies in Haemostasis and Thrombosis Associated with Liver Disease: Proceedings of the 7th International Coagulation in Liver Disease Conference. Thromb Haemost. 2018 Aug;118(8):1491-1506. doi: 10.1055/s-0038-1666861. Epub 2018 Jul 30. No abstract available. PMID 30060258
- [Result] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Result] Fan BE, Chong VCL, Chan SSW, Lim GH, Lim KGE, Tan GB, Mucheli SS, Kuperan P, Ong KH. Hematologic parameters in patients with COVID-19 infection. Am J Hematol. 2020 Jun;95(6):E131-E134. doi: 10.1002/ajh.25774. Epub 2020 Mar 19. No abstract available. PMID 32129508
- [Result] Cohen AT, Davidson BL, Gallus AS, Lassen MR, Prins MH, Tomkowski W, Turpie AG, Egberts JF, Lensing AW; ARTEMIS Investigators. Efficacy and safety of fondaparinux for the prevention of venous thromboembolism in older acute medical patients: randomised placebo controlled trial. BMJ. 2006 Feb 11;332(7537):325-9. doi: 10.1136/bmj.38733.466748.7C. Epub 2006 Jan 26. PMID 16439370
- [Result] Kumar M, Ahmad J, Maiwall R, Choudhury A, Bajpai M, Mitra LG, Saluja V, Mohan Agarwal P, Bihari C, Shasthry SM, Jindal A, Bhardwaj A, Kumar G, Sarin SK. Thromboelastography-Guided Blood Component Use in Patients With Cirrhosis With Nonvariceal Bleeding: A Randomized Controlled Trial. Hepatology. 2020 Jan;71(1):235-246. doi: 10.1002/hep.30794. Epub 2019 Aug 27. PMID 31148204
- [Derived] Premkumar M, Loganathan S, Kajal K, Hazarika A, Soni S, Puri GD, Sehgal IS, Suri V, Malhotra P, Singh V, Duseja A, Bhalla A, Ahluwalia J, Kumar N, Kekan K, Ram S, Singla K, Mahajan V, Yaddanapudi N. COVID-19-related dynamic coagulation disturbances and anticoagulation strategies using conventional D-dimer and point-of-care Sonoclot tests: a prospective cohort study. BMJ Open. 2022 May 2;12(5):e051971. doi: 10.1136/bmjopen-2021-051971. PMID 35501097